CLINICAL TRIAL: NCT00604084
Title: Veron Scabies Education and Eradication Program
Acronym: VSEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#2007/006
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Scabies
Keywords: Scabies; Ivermectin; Lindane; Mass Eradication
MeSH Terms: conditions — Scabies | interventions — Ivermectin; Permethrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivermectin (Experimental): Non-pregnant, non-breastfeeding, taller than 90cm and 5 years or older
  Interventions: Drug: Ivermectin
- Permethrin (Experimental): Pregnant, breastfeeding, children under 90cm or under 5 years old
  Interventions: Drug: Permethrin 5% lotion

INTERVENTIONS:
Drug: Ivermectin — Ivermectin 200ug/kg, 1 dose Q 6 months x 2, total duration = 12 months
  Other Names: Ivermectina
  Arms: Ivermectin
Drug: Permethrin 5% lotion — apply lotion to entire body, excluding head, at bedtime, rinse off following morning, wait one week, repeat application for a total of 2 applications, PRN frequency, NMT 6 applications in 12 months, total duration = 12 months.
  Other Names: Permethrina locion
  Arms: Permethrin

SUMMARY:
The purpose of this project is to develop a community scabies eradication and education program for the highly endemic areas surrounding the Veron community on the eastern tip of the Dominican Republic. It proposes the use of oral Ivermectin as a replacement for topical Lindane--a readily available medical formulation, pesticide, and environmental toxin that is reported to be banned in the Dominican Republic as well as over 80 other countries throughout the world.

DETAILED DESCRIPTION:
Introduction

The Secretaría de Estado de Salud Pública y Asistencia Social public health clinic in Veron, Dominican Republic continually reports a subjectively high prevalence and incidence of scabies infections among its general patient population without any means of direct measurement, proper intervention, or control, raising concerns that long-term infestation may lead to multiple other secondary medical and environmental problems.

The purpose of this project is to develop a community scabies eradication and education program for the highly endemic areas surrounding the Veron community. It proposes the use of oral Ivermectin as a replacement for topical Lindane, a readily available and prescribed pesticide and environmental toxin that is reportedly banned for all uses in the Dominican Republic as well as over 80 other countries throughout the world (Boffa, Brough, & Ead, 1995; Davies, Dedhia, Mergade, Banquet, & Maibach, 1983).

Ivermectin, on the other hand, is a remarkably safe, effective, cost-comparative oral medication with a substantially broader scope of coverage, duration of effectiveness, and ease of delivery and compliance when compared to Lindane, as well as over 20 years of use in global mass eradication campaigns for other parasites on the order of more than 50 million doses to date (Alexander, Bockarie, Kastens, Kazra, & Alpers, 1998; del Guidice, Chosidow, & Caumes, 2003; Madan, Jaskiran, Gupta, & Gupta, 2001).

Specific program goals include: the quantification of community disease prevalence, a statistically significant reduction in both scabies incidence as well as secondary disease sequelae, improved community scabies awareness and prevention abilities, and decreased environmental impact on the Veron area by eliminating the use of Lindane for scabies treatment.

The research is designed to employ a door-to-door survey and treatment campaign in a typical Veron neighborhood aimed at evaluating and treating every member in this target population to create a mass prophylaxis that breaks the parasite-host cycle. Another round of treatment will occur 6 months later, per pharmacologic dosage interval recommendations (del Guidice et al., 2003).

Individual and group scabies education programs will occur at the Veron clinic, as well as at the local schools to target the highly susceptible youth populations throughout the Veron area.

Incidence measurements will occur on a monthly basis for one year after program start, coinciding with two 6-month treatment intervals. At the end of one year, final scabies prevalence and incidence data will be evaluated for statistical significance. While mass treatments will cease at this time, oral Ivermectin will become the standard of care for ectoparasite coverage at the Veron clinic assuming a statistically significant reduction in scabies prevalence is achieved.

To date, no mass scabies eradication programs using oral Ivermectin have been reported in the Caribbean, despite it remarkable success in other countries against scabies as well as other parasites, namely onchocerciasis and filariasis (Walker & Johnstone, 2000; Walton & Holt, 2004). This project has the potential to be an important contribution to the effort to eradicate a source of significant morbidity for both the people of Veron and the global community as a whole.

Methodology

The Veron Scabies Eradication and Education Program will obtain all its priority population data via door-to-door interviews within the Barrio Nuevo neighborhood.

A survey team of medical personnel will walk door-to-door program in an attempt to survey and treat every inhabitant of Barrio Nuevo, unless there is refusal or absolute contraindications. Subjects will first be informed of the program and its intent, asked to sign a letter of patient confidentiality, and assigned a number identifier for tracking purposes.

After consent is obtained, a survey will be administered to collect basic demographic information, scabies knowledge indicators, as well as pertinent past and current medical history related to scabies infection and contraindications to treatment with Ivermectin.

The subject will then be asked to undergo a brief skin exam that assesses scabies infectivity and results recorded using the following criteria: the presence of erythematous popular, vesicular, pustular, or bullous lesions associated with itching. Information will be recorded and used to guide treatment protocol.

After the skin exam, subjects will be instructed on scabies medical treatment and prevention, given a patient information and education pamphlet, asked if they have any specific questions or concerns, informed of ongoing community scabies education workshops at the clinic, and instructed to return to the clinic in 2 weeks if they have an active scabies infection. Otherwise, they will be informed that the researchers will return to their neighborhood each month to collect more information and in 6 months to administer another treatment.

Finally, the subject will be given 200μg/kg oral Ivermectin dosed by height if they are male or non-pregnant/non-lactating female, 5 years of age or older, and taller than 90 cm.

If the subject is a female and of childbearing age (still menstruating on a monthly basis), not currently menstruating, not able to show proof of using oral contraceptives (birth control pills) or injectable contraceptives (scheduled Depo Provera), not surgically sterile (hysterectomy or tubal ligation) they will be asked to undergo a rapid urine pregnancy test. If the test is negative they will be given 200μg/kg oral Ivermectin dosed by height.

If the subject is knowingly pregnant or lactating, the rapid pregnancy test is positive, or a child under 5 years and shorter than 90 cm they will be instructed on how to properly use Permethrin 5% lotion and given a 60gm bottle.

This protocol will be followed until every household is visited and treated within Barrio Nuevo at time = 0 and again at time = 6 months.

Investigators will conduct monthly scabies incidence surveys via door-to-door skin checks within Barrio Nuevo looking for current scabies symptomatology and recording results on the form described above.

At the end of one year, final scabies prevalence and incidence data will be evaluated for statistical significance. While mass treatments will cease at this time, oral Ivermectin will become the standard of care for ectoparasite coverage at the Veron clinic assuming a statistically significant reduction in scabies prevalence is achieved.

ELIGIBILITY:
Inclusion Criteria:

IVERMECTIN ARM:

* able to swallow pills
* no known allergy to Ivermectin
* not pregnant
* not breastfeeding
* 5 years or older
* taller than 90cm
* willingness to participate in study and give written consent

PERMETHRIN ARM:

* no known allergy to Permethrin 5% lotion
* able to apply lotion to self or to other person if a child
* pregnant
* breastfeeding
* younger than 5 years
* shorter than 90cm
* willingness to participate in study and give written consent

Exclusion Criteria:

IVERMECTIN ARM:

* unable to swallow pills
* allergy to Ivermectin
* pregnant
* breastfeeding
* younger than 5 years
* shorter than 90cm
* unwilling to participate in study or give written consent

PERMETHRIN ARM:

* unable to apply lotion to self
* allergy to Permethrin 5% lotion
* not pregnant
* not breastfeeding
* 5 years or older
* taller than 90cm
* unwilling to participate in study or give written consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Scabies incidence | monthly

SECONDARY OUTCOMES:
Scabies-induced skin abscess incidence | monthly
Incidence of Lindane prescription and use | monthly
Incidence of Ivermectin prescription and use | monthly
Scabies disease, treatment, and prevention awareness | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy J White, DO, Principal Investigator — Virginia College of Osteopathic Medicine; Dean Sutphin, PhD, Study Chair — Virginia College of Osteopathic Medicine
Locations (1):
- Barrio Nuevo, Veron, La Altagracia Province, Dominican Republic

REFERENCES:
- [Background] Boffa MJ, Brough PA, Ead RD. Lindane neurotoxicity. Br J Dermatol. 1995 Dec;133(6):1013. doi: 10.1111/j.1365-2133.1995.tb06950.x. No abstract available. PMID 8547026
- [Background] Davies JE, Dedhia HV, Morgade C, Barquet A, Maibach HI. Lindane poisonings. Arch Dermatol. 1983 Feb;119(2):142-4. doi: 10.1001/archderm.1983.01650260050017. PMID 6186202
- [Background] Alexander ND, Bockarie MJ, Kastens WA, Kazura JW, Alpers MP. Absence of ivermectin-associated excess deaths. Trans R Soc Trop Med Hyg. 1998 May-Jun;92(3):342. doi: 10.1016/s0035-9203(98)91035-5. No abstract available. PMID 9861413
- [Background] del Giudice P, Chosidow O, Caumes E. Ivermectin in dermatology. J Drugs Dermatol. 2003 Jan;2(1):13-21. PMID 12852376
- [Background] Madan V, Jaskiran K, Gupta U, Gupta DK. Oral ivermectin in scabies patients: a comparison with 1% topical lindane lotion. J Dermatol. 2001 Sep;28(9):481-4. doi: 10.1111/j.1346-8138.2001.tb00015.x. PMID 11603388
- [Background] Walker GJ, Johnstone PW. Interventions for treating scabies. Cochrane Database Syst Rev. 2000;(3):CD000320. doi: 10.1002/14651858.CD000320. PMID 10908470
- [Background] Walton SF, Holt DC, Currie BJ, Kemp DJ. Scabies: new future for a neglected disease. Adv Parasitol. 2004;57:309-76. doi: 10.1016/S0065-308X(04)57005-7. PMID 15504541